CLINICAL TRIAL: NCT00781183
Title: Does Pulmonary Rehabilitation Change The Self-Selected And Maximum Sustainable Walking Speed In Patients With Symptomatic Lung Disease?
Brief Title: Does Pulmonary Rehabilitation Change Self-Selected And Maximum Sustainable Walking Speed In Patients With Lung Disease?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Directory Respiratory Medicine, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D6255L00002
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: COPD; Chronic Lung Disease
Keywords: COPD; rehabilitation; walking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulmonary rehabilitation (Experimental): patients that are enrolled in pulmonary rehabilitation
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — 6-weeks of in-patient pulmonary rehabilitation or 12-weeks of out-patient pulmonary rehabilitation

SUMMARY:
Exercise training has been shown to reduce breathlessness and improve the exercise tolerance of people with lung disease. However, the effect of exercise training on the walking speed selected by these people during day-to-day life is unknown. Furthermore,the investigator do not know if exercise training changes the maximum speed that these people can walk at for a long period of time. This study will examine the relationship between walking speed and walking endurance before and following exercise training in people with lung disease and contribute importantly to our understanding of how patients choose to walk in relation to their capabilities.

DETAILED DESCRIPTION:
Rationale: Pulmonary rehabilitation (PR) is considered a standard of care for patients with symptomatic lung disease. It has achieved strong evidence for reducing symptoms and improving exercise tolerance. Walking is the most common form of physical activity and most individuals need to walk in the course of their daily activities. Chosen walking speed is a good indicator of the debilitating effects of disease and improvement in usual walk speed has been associated with a substantial reduction in mortality in elderly subjects. Therefore, it is important for clinicians to understand how patients choose to walk in relation to their capabilities as well as to know how this relationship changes with PR.

The main purpose of this study is to examine the relationship between walking speed and walking endurance before and after PR.

Primary aim: to estimate the maximum walking speed that can be sustained for > 24 min (i.e. maximum sustainable walking speed; MSWS) from the relationship between walking speed and walking time in patients with symptomatic lung disease.

Secondary aims: (i) to determine if chosen speed during the endurance walk test is different from the MSWS, (ii) to determine if MSWS and speed chosen for the endurance walk test changes in response to PR and, (iii) to measure the repeatability of endurance walk time (EWT), defined as the duration a patient can walk at a self-selected pace before that first need to stop and rest.

Significance: Walking is the most common form of physical activity. Chosen walking speed and the capacity to endure walking at different speeds can help quantify disability. Also, studies that examine the effect of PR on survival are not available. However, indirect evidence suggests that PR improves many of the risk factors associated with mortality in patients with COPD. This study will examine the effect of PR on the usual walking speed selected by individuals with symptomatic lung disease, which has been demonstrated to be a predictor of mortality in elderly individuals. Therefore, our study may contribute to the indirect evidence for the effects of PR on survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to pulmonary rehabilitation with symptomatic chronic lung disease

Exclusion Criteria:

* Co-morbid conditions that adversely affect exercise capacity or participation in a pulmonary rehabilitation program; inability to provide written informed consent; weaning doses of oral corticosteroids or methylxanthines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Endurance walk time (EWT) defined as the time a patient can walk at a self-selected speed until they first need to stop and rest | Pre and post pulmonary rehabilitation
The maximum sustainable walk speed (MSWS) defined as the maximum speed that a patient walk for at for > 24 minutes | Pre and post pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dolmage TE, Evans RA, Hill K, Blouin M, Brooks D, Goldstein RS. The effect of pulmonary rehabilitation on critical walk speed in patients with COPD: a comparison with self-paced walks. Chest. 2012 Feb;141(2):413-419. doi: 10.1378/chest.11-1059. Epub 2011 Jul 21. PMID 21778262
- [Derived] Evans RA, Hill K, Dolmage TE, Blouin M, O'Hoski S, Brooks D, Goldstein RS. Properties of self-paced walking in chronic respiratory disease: a patient goal-oriented assessment. Chest. 2011 Sep;140(3):737-743. doi: 10.1378/chest.10-3104. Epub 2011 Mar 10. PMID 21393393